CLINICAL TRIAL: NCT02745028
Title: Effect of a Single Dose of Monosodium Glutamate on Delayed Gastric Emptying in Children
Brief Title: Monosodium Glutamate on Gastric Emptying
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol was cancelled becouse lack of funding
Sponsor: Veronica Beatriz Busoni (Other)
Collaborators: International Glutamate Technical Committee (Unknown)
Responsible Party: Sponsor-Investigator, Veronica Beatriz Busoni, Head of the Pediatric Gastroenterology and Hepatology Service, Hospital Italiano de Buenos Aires
Organization: Hospital Italiano de Buenos Aires (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2404
Record Dates: First submitted 2016-04-07; First posted 2016-04-20 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Delayed Gastric Emptying
Keywords: delayed gastric emptying; children; monosodium glutamate
MeSH Terms: conditions — Gastroparesis | interventions — Sodium Glutamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- With monosodium glutamate (Other): Results of one time gastric emptying study with a single dose of monosodium glutamate; 1 g for weight greater than 45 kg, 700mg between 35 and 44,900 kg, 600mg between 25 and 34,900, 500mg between 15 and 25 kg and 250mg in less than 15 kg
  Interventions: Dietary Supplement: Monosodium glutamate

INTERVENTIONS:
Dietary Supplement: Monosodium glutamate — A single dose of weight adjusted monosodium glutamate will be added at the time of a repeat radionuclide gastric emptying study

SUMMARY:
Children with a radionuclide gastric emptying test with abnormal results will undergo a second test with the addition of a weight adjusted dose of monosodium glutamate. The purpose of the study is to determine if a single dose of monosodium glutamate can shorten the gastric emptying time.

DETAILED DESCRIPTION:
There is evidence that monosodium glutamate has effects on synapsis at the gastric and duodenum level that results in stimulation of contractility resulting on increase rate of gastric emptying. The purpose of the study is to demonstrate that the administration of a single dose of monosodium glutamate can shorten the gastric emptying time.

Patients with a prior study indicating a delay of gastric empting time, will undergo a second test with the addition of a weight adjusted dose of monosodium glutamate. Each patient will serve as her/his own control. Results will be analysed by pair-T test.

ELIGIBILITY:
Inclusion Criteria:

* children with delayed gastric emptying not receiving prokinetic medication in the last 72 hours

Exclusion Criteria:

* Prior gastrointestinal surgery, patients with known history of reaction to monosodium glutamate. History of neoplasia, autoimmune or inflammatory bowel disease.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Reduced gastric emptying time | During the test (4 hours from intake)
  Percentage of reduction of gastric emptying time when glutamate is administered compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Veronica B Busoni, MD, Principal Investigator — Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Teramoto H, Shimizu T, Yogo H, Nishimiya Y, Hori S, Kosugi T, Nakayama S. Gastric emptying and duodenal motility upon intake of a liquid meal with monosodium glutamate in healthy subjects. Physiol Rep. 2014 Jan 6;2(1):e00187. doi: 10.1002/phy2.187. eCollection 2014 Jan 1. PMID 24744869
- [Result] Zai H, Kusano M, Hosaka H, Shimoyama Y, Nagoshi A, Maeda M, Kawamura O, Mori M. Monosodium L-glutamate added to a high-energy, high-protein liquid diet promotes gastric emptying. Am J Clin Nutr. 2009 Jan;89(1):431-5. doi: 10.3945/ajcn.2008.26180. Epub 2008 Dec 3. PMID 19056566
- [Result] Boutry C, Matsumoto H, Airinei G, Benamouzig R, Tome D, Blachier F, Bos C. Monosodium glutamate raises antral distension and plasma amino acid after a standard meal in humans. Am J Physiol Gastrointest Liver Physiol. 2011 Jan;300(1):G137-45. doi: 10.1152/ajpgi.00299.2010. Epub 2010 Oct 28. PMID 21030612
- [Result] Hosaka H, Kusano M, Zai H, Kawada A, Kuribayashi S, Shimoyama Y, Nagoshi A, Maeda M, Kawamura O, Mori M. Monosodium glutamate stimulates secretion of glucagon-like peptide-1 and reduces postprandial glucose after a lipid-containing meal. Aliment Pharmacol Ther. 2012 Nov;36(9):895-903. doi: 10.1111/apt.12050. PMID 22978669
- See also: Questions and Answers on Monosodium glutamate — http://www.fda.gov/food/ingredientspackaginglabeling/foodadditivesingredients/ucm328728.htm